CLINICAL TRIAL: NCT03896672
Title: How To Use Non-Invasive Positive Airway Pressure In Pleural Effusion Drainage: Protocol For Implementation Multicentric Scientific Evidence With Audit
Brief Title: Clinical Implementation of the Use of Positive Pressure in Chest Drainage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Adriana Claudia Lunardi, Principal Investigator, Universidade Cidade de Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UNIFAP
Record Dates: First submitted 2019-03-15; First posted 2019-04-01 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Pleural Effusion
Keywords: Clinical Practice Based on Scientific Evidence; Non-Invasive Positive Airway Pressure; Pleural effusion; Chest drain; Physical therapy
MeSH Terms: conditions — Pleural Effusion | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with Continuous Positive Airway Pressure (Experimental): All patients will undergo to physiotherapeutic treatment based on the previous training of the physiotherapist
  Interventions: Device: Continuous Positive Airway Pressure

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — Continuous Positive Airway Pressure will be applied three times daily during 7 consecutive days, if the physiotherapist follow the previous training. Each application should during 30 minutes. Pressure should be adjusted in 15 centimeters of water.

SUMMARY:
Background: Scientific evidence appoints that the use of non-invasive positive airway pressure in pleural effusion drainage patients is associated with a reduction in these complications, as well as with other benefits. Objectives: To test the implementation of the best evidence-based practices for the use of non-invasive continuous positive airway pressure (CPAP) in patients with chest drainage for pleural effusion, by acceptability, reach, appropriateness, direct costs, feasibility, fidelity, penetration, and sustainability. In addition, to assess the impact of implementing these practices on health-related outcomes of patients having their pleural effusion drained through dwelling time of the chest tube, hospital stay and others relevant outcomes. Methods: quasi-experimental study with pretest-posttest design. Eight hospitals that provide physiotherapeutic care to pleural effusion drainage patients will be involved. The study will be developed in three phases. In phase I, a audit team will help the local research team to elaborate strategies to cope with barriers related to the use of CPAP in patients with pleural effusion and catheter drainage, using a interview with the physical therapist, patient history analysis, and interviews with the patients. In implementation phase, the results obtained from phase I will be presented to physiotherapists to physiotherapists and a discussion will be started on the evidence regarding the best practices in the application of CPAP for educational purposes only. In phase III, new interviews will be held with the physical therapist and patients and the patient histories will be analyzed to assess the impact of the intervention 30 days after implementation phase.

DETAILED DESCRIPTION:
Design: Effectiveness-implementation hybrid designs, type 3 (primary focus on implementation; secondary focus on effectiveness).

Study setting and Participants: Seven hospitals in Brazil and one in Belgium will be included in the study. The investigators will invite physical therapists working in sectors where patients with pleural effusion and chest tube are hospitalized and the patients themselves to participate in this study.

Study design: The study will be developed in three phases:

* Pre-audit and baseline audit (Phase I)
* Transfer of best practices (Phase II)
* Post-intervention audit (Phase III) a. Pre-audit and baseline audit phase: the purpose of this phase will be to establish the audit team that will discuss the inclusion of health professionals and patients in the study. The audit team will be composed of two local members selected from researchers, clinical director, administrative director, technical director, coordinator, or head of physiotherapy/rehabilitation unit-department in each hospital. As a way to increase physical therapists' participation, the audit team of each hospital will be responsible for the intervention (Phase II - Transfer phase of best practices).

The audit team will check the current local physiotherapeutic practices in the use of Continuous Positive Airway Pressure (CPAP) in patients with pleural effusion drainage exclusively based on scientific evidence and evaluation of the feasibility of measuring the proposed outcomes. In addition, the team will try to identify the possible barriers to be faced in previously scheduled meetings, for example, institutional routines and availability of resources. This audit team can help the research team to develop strategies for coping with these barriers through a structured interview with physical therapists (including questions regarding sociodemographic issues, use of CPAP therapy, physiotherapeutic visits, number of visits and physiotherapeutic techniques) as well as with pleural effusion patients (including questions on the use of therapies applied by the physical therapist, number of daily physiotherapeutic visits, level of tolerance to the use of CPAP, level of satisfaction with physical therapy and level of pain) or by another feasible form discussed at the time. The collection of information from the physiotherapists, patients and medical records simultaneously aims to verify the consistency of the information and the measuring of the outcomes prior to the intervention through historical control.

Audit criteria:

Previously established criteria listed below:

1. Increase in: adherence, adoption, appropriateness, fidelity, tolerability of non-invasive positive pressure treatment, and level of participant satisfaction with treatment.
2. Reduction in: dwelling time of thoracic tube, length of hospital stay, pulmonary complication rate, need for antibiotic therapy, treatment costs, pain level of the patient before and immediately after treatment, and adverse effects.

Baseline evaluation of outcomes and physiotherapeutic practices with CPAP use in patients with pleural effusion and chest tube:

Before the transfer of best practices (Phase II), the outcomes of interest established in the audit criteria will be discussed and confirmed by the audit team, and the clinical practices used by the physical therapist will be identified through interviews, as well as the patients' reports.

In order to assess the efficiency of the implementation process, medical records of patients included in this study will be compared to a historical cohort, i.e. medical records of patients with PE that have been hospitalized in the previous 6 months will be retrieved and compared.

The following information will be collected from the patient medical records:

* Tolerability of CPAP treatment
* Dwelling time of thoracic tube
* Length of hospital stay
* Presence of pulmonary complication
* Use of antibiotics therapy
* Estimate of treatment costs (information that can help in the estimation of costs are, among others: materials and medicines used, hotel, length of stay)
* Presence of adverse effects (aerophagia and pleural or bronchopleural fistula)
* Number of physiotherapy sessions
* Physiotherapy techniques applied to patients

  b. Transfer phase of best practices: will also be called the intervention phase. This phase will present to the physical therapists the results extracted from phase I, besides raising a discussion on the best evidence available with mere educational goals. For this intervention, educational materials (seminars, posters, and newsletters), educational outreach activities (interactive face-to-face instruction, workshops, roundtable, and discussion committee), reminders (posters, stickers, and buttons) and messages by electronic media will be used, during an event with the same approaches for each hospital, i.e. continuing education. All approaches will be carried out as homogeneously as possible in all hospital settings to minimize bias.

A full CPAP kit (Müller Resuscitator, Engesp, Brazil) will be donated to each hospital if it is not available onsite. Each kit contains 1 injector, 1 vaporizer, 1 "T" connection, 1 manual valve, 1 oxygen pressure regulator, 2 face masks for inhalation with inflatable cushion, 1 head attachment gear for the mask. In addition, training will be offered on the use of the device.

c. Post-intervention audit phase: all the criteria for inclusion will be maintained in this phase and a new interview will be held with the same physical therapists and patients that have been involved in phase I. Furthermore, medical records of patients and the historical cohort will be analyzed and compared to evaluate the impact of the intervention. This phase will take place 30 days after the end of the second phase, based on a recent study13. In addition, in another study, it was also suggested that this phase can also be started 30 days after the end of the second phase14.

The new structured interview with the physical therapists will occur only once in each phase I and phase III, through a structured form face-to-face or by other communication media, such as email, telephone, or any other means that is convenient for the professional. This will take place in the hospital, office, home or other place and time at the physical therapist's convenience.

The interview with the patients (who have already received or are receiving physical therapy, in order to check what has been done in their physiotherapeutic treatment) will be held by means of a structured form, face-to-face or using other communication media, such as e-mail, telephone, or any other means that is convenient for the patient. The interview will be applied at three different moments. First, within 24 hours after the insertion of chest drain in the hospital. Second, between 10 and 12 days after the drainage tube has been inserted (please correct if I am wrong) and only for the variables infection and pain level. Third, 30 days after the drainage. The two latter interviews will take place in the hospital, office, home or other place and time at the patient's convenience.

ELIGIBILITY:
Inclusion Criteria for professionals:

- Graduated physical therapists working in the sectors where patients with PE and chest drainage are hospitalized.

Inclusion Criteria for patients:

* 18 years or older
* with pleural effusion diagnosed by the physician
* undergo to chest drainage less than 24 hours earlier

Exclusion Criteria for professionals:

- Physical therapists taking internships in these hospitals and physical therapists who fail to participate in at least one phase of the study will be excluded.

Exclusion Criteria for patients:

- contraindications for the use of CPAP (such as drowsiness, restlessness, treatment refusal, hemodynamic instability, systolic blood pressure <90 mmHg, facial trauma, ineffective cough or swallowing impairment, vomiting, upper gastrointestinal bleeding, acute myocardial infarction in the past 48 hours or bullous emphysema).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Rate of adherence to treatment by patients and by professionals | through study completion, an average of 1 years
  Adherence will be assessed by the level of satisfaction of the treatment with CPAP use among the participants (patients and professionals).
Rate of appropriateness of the treatment according to previous professional training | through study completion, an average of 1 years
  Appropriateness will be evaluated through the perception of physical therapist about the adequacy of the use of CPAP for the treatment of patients with PE drained in the hospital environment.
Treatment direct costs | through study completion, an average of 1 years
  Treatment costs will be estimated based on the informed daily hospital fees, antibiotics use, physiotherapy session, equipment and accessories for the use of CPAP during the hospitalization period of each patient.
Rate of treatment feasibility | through study completion, an average of 1 years
  Feasibility will be evaluated through the success or unsuccess of the use of noninvasive positive pressure in the treatment of drainage drainage within the hospital environment. Successful viability will be determined if there is a decrease in adverse effects, pulmonary complications, and need for antibiotics, and increased tolerance of CPAP use.
Penetration of professional training | through study completion, an average of 1 years
  Service access the integration of the use of CPAP in the treatment of chest drained for pleural effusion within the hospital service and its subsystems will be assessed by the following operation: Total number of people with any contact with the service during the year (number of eligible persons who use a service), divided by Total eligible persons at some point during the year (total number of persons eligible for the service)14. This penetration (annual penetration) is the most used in research because it is very easy to perform
Rate of sustainability of professional training | through study completion, an average of 1 years
  Sustainability will be assessed by the Level of Institutionalization scales for health promotion programs proposed by Goodman et al.

SECONDARY OUTCOMES:
Chest drainage duration | through study completion, an average of 1 years
  The number of days of the chest drainage will be recorded
Hospitalization duration | through study completion, an average of 1 years
  The days of hospitalization after the chest drainage until the hospital discharge of each patient will be recorded
Rate of pulmonary complications | through study completion, an average of 1 years
  the complications considered will be: pneumonia, atelectasis, or lung entrapment. These complications will be recorded based on clinical, laboratory and imaging exams up to the hospital discharge
Rate of adverse effects | through study completion, an average of 1 years
  the adverse effects for the use of noninvasive positive pressure considered will be aerophagia and bronchopleural fistula. These adverse effects will be recorded until the hospital discharge
Rate of need for antibiotics therapy | through study completion, an average of 1 years
  Need for antibiotics therapy: it will be registered based on the medical prescription on the 1st day of hospitalization, between 3 and 4 days, between 10 and 12 days, and 30 days after the chest drainage
Level of tolerance of noninvasive positive pressure use | through study completion, an average of 1 years
  tolerance will be assessed using the visual analog scale from zero to ten, zero corresponding to fully tolerable (no discomfort) and ten to totally intolerable (unbearable discomfort).
Pain level of the patient: visual analog scale | through study completion, an average of 1 years
  the pain level of the patient will be assessed using the visual analogic scale ranging from zero to ten, where zero equals the total absence of pain and ten equals unbearable pain, during the patient's inclusion, between 10 and 12 days, and 30 days after the chest drainage

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Lunardi, PhD, Principal Investigator — Universidade Cidade de São Paulo
Locations (1):
- Hospital das Clínicas Dr. Alberto Lima, Macapá, Amapá, Brazil

REFERENCES:
- [Background] Medford AR, Maskell N. Pleural effusion. Postgrad Med J. 2005 Nov;81(961):702-10. doi: 10.1136/pgmj.2005.035352. PMID 16272233
- [Background] Krishna R, Antoine MH, Alahmadi MH, Rudrappa M. Pleural Effusion. 2024 Aug 31. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK448189/ PMID 28846252
- [Background] Maskell N; British Thoracic Society Pleural Disease Guideline Group. British Thoracic Society Pleural Disease Guidelines--2010 update. Thorax. 2010 Aug;65(8):667-9. doi: 10.1136/thx.2010.140236. No abstract available. PMID 20685739
- [Background] McDermott S, Levis DA, Arellano RS. Chest drainage. Semin Intervent Radiol. 2012 Dec;29(4):247-55. doi: 10.1055/s-0032-1330058. PMID 24293797
- [Background] Oliveira JF, Mello FC, Rodrigues RS, Boechat AL, Conde MB, Menezes SL. Effect of continuous positive airway pressure on fluid absorption among patients with pleural effusion due to tuberculosis. Rev Bras Fisioter. 2010 Mar-Apr;14(2):127-32. doi: 10.1590/s1413-35552010005000001. Epub 2010 Apr 30. PMID 20464170
- [Background] da Conceicao Dos Santos E, Lunardi AC. Efficacy of the addition of positive airway pressure to conventional chest physiotherapy in resolution of pleural effusion after drainage: protocol for a randomised controlled trial. J Physiother. 2015 Apr;61(2):93. doi: 10.1016/j.jphys.2014.11.016. Epub 2015 Mar 3. PMID 25744852
- [Background] Nedjat S, Gholami J, Yazdizadeh B, Nedjat S, Maleki K, Majdzadeh R. Research's Practice and Barriers of Knowledge Translation in Iran. Iran J Public Health. 2014 Jul;43(7):968-80. PMID 25909064
- [Background] Karin H, Filip S, Jo G, Bert A. Obstacles to the implementation of evidence-based physiotherapy in practice: a focus group-based study in Belgium (Flanders). Physiother Theory Pract. 2009 Oct;25(7):476-88. doi: 10.3109/09593980802661949. PMID 19925170
- [Background] Schettino GP, Reis MA, Galas F, Park M, Franca SA, Okamoto VN, Carvalho CR. [Noninvasive mechanical ventilation with positive pressure]. Rev Bras Ter Intensiva. 2007 Jun;19(2):245-57. Portuguese. PMID 25310789
- [Background] Cortes CT, Santos RC, Caroci Ade S, Oliveira SG, Oliveira SM, Riesco ML. [Implementation methodology of practices based on scientific evidence for assistance in natural delivery: a pilot study]. Rev Esc Enferm USP. 2015 Oct;49(5):716-25. doi: 10.1590/S0080-623420150000500002. Portuguese. PMID 26516739
- [Background] Stiles PG, Boothroyd RA, Snyder K, Zong X. Service penetration by persons with severe mental illness: how should it be measured? J Behav Health Serv Res. 2002 May;29(2):198-207. doi: 10.1007/BF02287706. PMID 12032977
- [Background] Steckler A, Goodman RM, McLeroy KR, Davis S, Koch G. Measuring the diffusion of innovative health promotion programs. Am J Health Promot. 1992 Jan-Feb;6(3):214-24. doi: 10.4278/0890-1171-6.3.214. PMID 10148679
- [Background] Goodman RM, McLeroy KR, Steckler AB, Hoyle RH. Development of level of institutionalization scales for health promotion programs. Health Educ Q. 1993 Summer;20(2):161-78. doi: 10.1177/109019819302000208. PMID 8491630
- [Background] Scheirer MA, Dearing JW. An agenda for research on the sustainability of public health programs. Am J Public Health. 2011 Nov;101(11):2059-67. doi: 10.2105/AJPH.2011.300193. Epub 2011 Sep 22. PMID 21940916
- [Background] Barab SA, Redman BK, Froman RD. Measurement characteristics of the levels of institutionalization scales: examining reliability and validity. J Nurs Meas. 1998 Summer;6(1):19-33. PMID 9769609
- [Background] Scurlock-Evans L, Upton P, Upton D. Evidence-based practice in physiotherapy: a systematic review of barriers, enablers and interventions. Physiotherapy. 2014 Sep;100(3):208-19. doi: 10.1016/j.physio.2014.03.001. Epub 2014 Mar 12. PMID 24780633
- [Background] Olsen NR, Bradley P, Lomborg K, Nortvedt MW. Evidence based practice in clinical physiotherapy education: a qualitative interpretive description. BMC Med Educ. 2013 Apr 11;13:52. doi: 10.1186/1472-6920-13-52. PMID 23578211